CLINICAL TRIAL: NCT05222139
Title: "Multicenter Observational Study to Assess the Incidence and Features of COVID-19 and the Response to COVID-19 Vaccination in Fragile Patients"
Brief Title: Monitoring COVID-19 Vaccination Response in Fragile Populations
Acronym: ORCHESTRA-4
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Collaborators: Universita di Verona (Other); Hospital Universitario Virgen Macarena (Other); Azienda Ospedaliera di Padova (Other); Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Ulss 2 Marca Trevigiana (Other); University College Dublin (Other); Luxembourg Institute of Health (Other Government); Fondazione ICONA (Other); University Medical Center Groningen (Other); University of Buenos Aires (Other); PENTA Foundation (Network); Universiteit Antwerpen (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Helmholtz Zentrum München (Industry); CINECA consorzio universitario italiano (Unknown); Charite University, Berlin, Germany (Other); Centre de Recherche Médicale de Lambaréné (Other)
Responsible Party: Principal Investigator, Maddalena Giannella, Professor, University of Bologna
Other Study IDs: ORCHESTRA-4
Record Dates: First submitted 2021-11-08; First posted 2022-02-03 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: SARS CoV 2 Infection; Vaccination; Infection; Breakthrough Infection
Keywords: Frail patients
MeSH Terms: conditions — COVID-19; Infections; Breakthrough Infections | interventions — heterologous prime boost COVID-19 vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biological samples (including blood, naso-pharingeal swabs, urine, and stool) will be collected and stored in the biobank of each participating center according to local authority regulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Solid organ transplant recipients: Solid organ transplant recipients
  Interventions: Biological: COVID-19 vaccination
- People living with HIV: People living with HIV
  Interventions: Biological: COVID-19 vaccination
- Patients with oncological diseases: Patients with oncological diseases
  Interventions: Biological: COVID-19 vaccination
- Patients with hematological diseases: Patients with hematological diseases
  Interventions: Biological: COVID-19 vaccination
- Patients with cystic fibrosis: Patients with cystic fibrosis
  Interventions: Biological: COVID-19 vaccination
- Patients with Parkinson Disease: Patients with Parkinson Disease
  Interventions: Biological: COVID-19 vaccination
- Patients with rheumatological diseases: Patients with rheumatological diseases
  Interventions: Biological: COVID-19 vaccination
- Pregnant women/ New-borns: Pregnant women/ New-borns
  Interventions: Biological: COVID-19 vaccination
- Children: Children
  Interventions: Biological: COVID-19 vaccination

INTERVENTIONS:
Biological: COVID-19 vaccination — Monitoring COVID-19 vaccination

SUMMARY:
The present study is part of ORCHESTRA project, a three-year international research project aimed at tackling the coronavirus pandemic. ORCHESTRA provides an innovative approach to learn from the pandemic SARS-CoV-2 crisis, derive recommendations to further management of COVID-19 and be prepared for the possible future pandemic waves. The ORCHESTRA project aims to deliver sound scientific evidence for the prevention and treatment of the infections caused by SARS-CoV-2 assessing epidemiological, clinical, microbiological, and genotypic aspects of population, environment and socio-economic features. The project builds upon existing, and new largescale population cohorts in Europe (France, Germany, Spain, Italy, Belgium, Romania, Netherlands, Luxemburg, and Slovakia) and non-European countries (India, Perú, Ecuador, Colombia, Venezuela, Argentina, Brazil and Gabon) including SARS-CoV-2 infected and non-infected individuals of all ages and conditions. The primary aim of ORCHESTRA is the creation of a new pan European cohort applying homogenous protocols for data collection, data sharing, sampling, and follow-up, which can rapidly advance the knowledge on the control and management of the COVID-19. ORCHESTRA will include SARS-CoV-2-negative individuals and thereby enable a prospective follow-up and an analysis of vaccination response. The cohort will involve four different populations: general population, COVID-19 patients, fragile individuals (children, elderly, transplanted, oncological, HIV infected, and those with Parkinson disease), and health-care workers. Each of these "perpetual" cohorts can answer different research questions and vaccine strategies.

Within the ORCHESTRA project, the Work Package 4 (WP4) will focus on the cohort of fragile patients including pregnant women/new-born, children, patients with HIV infection, patients with autoimmune disease, solid organ transplant recipients, patients with oncological and hematological diseases, patients with cystic fibrosis, patients with Parkinson Disease and rheumatological diseases from from 14 countries (5 European and 9 non-European countries), with approximately 20000 subjects.

DETAILED DESCRIPTION:
Since the beginning of COVID-19 pandemic, several special settings have been identified regarding the susceptibility to SARS-CoV-2 infection, the associated clinical spectrum and outcome. The participants include pregnant women, pediatric patients, elderly in particular those whole live in long-term care facilities (LTCFs), and immunocompromised hosts including solid organ transplant recipients (SOT), hematopoietic stem cell transplant (HSCT) recipients and patients with cancer. Among pregnant women and children, asymptomatic or mild diseases have been frequently reported, prompting controversial concerns about their role in the infection transmission in community and hospital settings.

On the other hand, a high impact of COVID-19 on morbidity and mortality has been described in elderly and immuno-compromised hosts. Thus, optimization of prevention strategies, screening practices and therapeutic management is strongly advocated in fragile patients. Indeed, these settings have been established as priority groups for vaccines. However, safety and efficacy of vaccination in these populations should be carefully assessed. Thus, preliminary epidemiological data are strongly needed to design further intervention trials and health policies.

Besides, an increasing body of evidence suggests that the gut microbiota plays a role in determining the severity of COVID-19, possibly through the modulation of immune responses. Furthermore, dysbiosis of the gut microbiota could contribute to the persistence of symptoms, even after the resolution of the disease.

For the same reasons, the microbiota could be involved in the onset of adverse reactions induced by vaccination, especially in fragile populations, as recently discussed. Defining the impact of the microbiota on immunity to vaccination and therefore on its effectiveness is currently considered a priority in various clinical settings.

Moreover, early observations show that vaccines do not induce an immune response conferring protection to many fragile patients, resulting in severe Covid-19 cases. It is important to understand what cellular networks and molecular pathways are switched on/off by the administration of vaccines, and to identify the biological patterns that characterize responders and non-responders. DNA methylation and gene expression analyses may inform on the genomic patterns involved in response to vaccines and in the differences between responders and non-responders. Indeed, DNA sequencing may reveal that the perturbation detected at the regulatory levels may be influenced by alterations in the genome of the divergent subjects.

With this premise, the Investigators deem that a WP dedicated to fragile patients in the ORCHESTRA project is necessary to inform about the peculiarities of the fragile cohort as a whole, and of each subgroup as well, providing clinical and biological information useful to design targeted prevention and therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Any age
* Any comorbidity
* Person (or attorney or deputy who has been authorized to make the decision for patients who lack capacity) consent to participate or appropriate local waiver of consent.

Exclusion Criteria:

* Patients did not agree to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all age and any comorbidity included in an ORCHESTRA fragile population cohort
Sampling Method: Probability Sample
Enrollment: 8894 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-07-16 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Early immune response to COVID-19 vaccine patients | 3 ± 1 month after vaccination onset
  To investigate the early immune response to COVID-19 vaccine in fragile patients assessing the levels of antibodies against Spike antigens and the patterns of cellular immune response
Late immune response to COVID-19 vaccine | 12 ± 3 months after vaccination onset
  To investigate the late immune response to COVID-19 vaccine in fragile patients assessing the levels of antibodies against Spike antigens and the patterns of cellular immune response
Rate of COVID-19 breakthrough infections | within 1 year after vaccination onset
  To investigate the rate of COVID-19 breakthrough infections in fragile patients within 1 year after vaccination onset
Rate of hospital admission for COVID-19 breakthrough infections condition and its impact on the outcome in fragile patients | within 1 year after vaccination onset
  To investigate the rate of hospital admission for COVID-19 breakthrough infections in fragile patients
Rate of death for COVID-19 breakthrough infections patients | within 1 year after vaccination onset
  To investigate the rate of death for COVID-19 breakthrough infections in fragile patients

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Giannella, MD PhD, Principal Investigator — University of Bologna
Locations (20):
- Universidad de Buenos Aires (UBA), Buenos Aires, Argentina
- Centre de Recherches Medicales de Lambaréné (CERMEL), Lambaréné, Gabon
- India (2):
  - Catholics Bishops Conference of India, Society for Medical Education (CBCI), Bangalore
  - Translational Health Science and Technology Institute (THSTI), Faridabad
- Italy (13):
  - University of Bologna, Bologna
  - ICONA Foundation, Milan
  - Aziena Ospedaliera Universitaria di Padova - Centro Trapianti di fegato, Padua
  - Azienda Ospedaliera Universitaria di Padova - Centro trapianti di polmone, Padua
  - Azienda Ospedaliera Universitaria di Padova - UOC Chirurgia dei trapianti di rene, Padua
  - Azienda Ospedaliera Universitaria di Padova - UOC Nefrologia Pediatrica, Padua
  - Azienda Ospedaliero Universitaria di Padova - Clinica Medica 5, Padua
  - Azienda Ospedaliero Universitaria di Padova - Trapianto Multiviscerale, Padua
  - Azienda Ospedaliero Universitaria di Padova - UOC Cardiochirurgia, Padua
  - Azienda Ospedaliero Universitaria di Padova - UOC Clinica Pediatrica, Padua
  - PENTA Foundation, Padua
  - Azienda ULSS2 Marca Trevigiana, Treviso
  - University of Verona, Verona
- Luxembourg Institute of Health (LIH), Luxembourg, Luxembourg
- University Medical Center Groningen (UMCG), Groningen, Netherlands
- Hosp. Univ. Virgen Macarena / Universidad de Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: SARS-CoV-2 vaccination in solid-organ transplant recipients: What the clinician needs to know. — https://pubmed.ncbi.nlm.nih.gov/34450686/
- See also: Evaluation of the kinetics of antibody response to COVID-19 vaccine in solid organ transplant recipients: the prospective, multicenter ORCHESTRA cohort. — https://pubmed.ncbi.nlm.nih.gov/35630462/
- See also: Relationship Between Immune Response to Severe Acute Respiratory Syndrome Coronavirus 2 Vaccines and Development of Breakthrough Infection in Solid Organ Transplant Recipients: The CONTRAST Cohort — https://pubmed.ncbi.nlm.nih.gov/36636955/
- See also: Effect of a Fourth Dose of mRNA Vaccine and of Immunosuppression in Preventing SARS-CoV-2 Breakthrough Infections in Heart Transplant Patients. — https://pubmed.ncbi.nlm.nih.gov/36985328/
- See also: Using machine learning to predict antibody response to SARS-CoV-2 vaccination in Solid Organ Transplant Recipients. The multicentre ORCHESTRA cohort. — https://pubmed.ncbi.nlm.nih.gov/37150358/
- See also: SARS-CoV-2 mRNA Vaccine Response in People Living with HIV According to CD4 Count and CD4/CD8 Ratio. — https://pubmed.ncbi.nlm.nih.gov/38005996/
- See also: SARS-CoV-2 mRNA vaccination and short-term changes in viral load and CD4/CD8 T-cell counts in people living with HIV — https://pubmed.ncbi.nlm.nih.gov/38643867/

DOCUMENTS (1):
  • Study Protocol (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT05222139/Prot_000.pdf